CLINICAL TRIAL: NCT06961084
Title: Comparison of I-124 PET/CT to I-123 Whole Body Imaging for the Diagnosis of Thyroid
Brief Title: Comparison of I-124 PET/CT for the Diagnosis of Thyroid Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Hope (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Thomas Hope, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 249212; NCI-2025-03041 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Thyroid Cancer
Keywords: Imaging Studies
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Iodine-124; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intervention: I-124 PET/CT (Experimental): All participants will be administered an oral dose of 60 to 85 megabecquerel (MBq) +/- 10% for I-124 (capsule) prior to the Positron Emission Tomography (PET) imaging. Scan coverage will extend from the vertex to the mid-thighs and in certain circumstances, coverage may be extended to the toes. Imaging will be acquired 20-28 hours after I-124 administered. Participants will be followed up for any adverse events for up to 5 days after the scan has been completed.
  Interventions: Drug: Iodine-124; Procedure: Positron Emission Tomography (PET)/Computerized tomography (CT)

INTERVENTIONS:
Drug: Iodine-124 — Given Orally
  Other Names: I-124; I-124 Radioisotope
Procedure: Positron Emission Tomography (PET)/Computerized tomography (CT) — Combination of PET and CT imaging
  Other Names: PET/CT

SUMMARY:
Persons diagnosed with thyroid cancer are often treated initially with a thyroidectomy, which is followed by ablation using Iodine-131, a therapy which has been shown to be effective and safe. Imaging of metastatic thyroid cancer has been performed with whole body I-131 and Iodine 123 (I-123) imaging for many decades and use I-123 for staging studies. Iodine 124 (I-124) is a radioisotope of iodine which emits a positron and is imaged using PET (positron emission tomography). This is a single arm prospective trial that evaluates the ability of Iodine-124 (I-124) to detect metastatic thyroid cancer compared to non-interventional, usual care I-123 and I-131 images.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1) Agreement between 1-124 PET and 1-123/1-131 SPECT.

SECONDARY OBJECTIVES:

1. Sensitivity and specificity of I-124 PET to detect metastatic thyroid cancer compared to composite standard.
2. Reclassification rate of I-124 PET compared to I-123 SPECT.
3. Inter-reader variability for I-124 PET and I-123 SPECT.
4. Safety of I-124 PET.
5. Participant level detection rate for I-124 in the overall population.
6. Participant level detection rate for I-124 in participants who have negative I-123 SPECT.
7. Comparison of lesion detection between I-124 PET and 24 hour I-123 SPECT.
8. Comparison of lesion detection between I-124 PET and post-treatment I-131 SPECT.

EXPLORATORY OBJECTIVES:

1. Ability to predict lesion absorbed dose using I-124 PET/CT.

OUTLINE:

All participants will have a single PET/CT scan after administration of I-124 and will be followed for up to 3-5 days by phone for evaluation of adverse events. A subset of participants being evaluated for dosimetry will be imaged up to two additional times over five days after administration. Data from other scans for comparison will be obtained from the participant's medical record.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years.
2. Histopathologically confirmed differentiated thyroid cancer, with clinical concern for metastatic disease:

   1. Metastatic disease seen on I-123 SPECT, Fluorodeoxyglucose (FDG) PET, CT scan or ultrasound.
   2. Elevated thyroglobulin in participant after total thyroidectomy.

   i. Participants with an undetectable thyroglobulin will be allowed if thyroglobulin antibodies are present.
3. Meeting criteria for one of the following two populations:

   1. American Thyroid Association (ATA) intermediate or high-risk thyroid cancer and planning on treatment using I-131.
   2. Metastatic disease on imaging (CT, MRI, ultrasound or FDG PET), and considering localized therapy such as surgery and radiation therapy.
4. Undergone total thyroidectomy.
5. Planned I-123 imaging within 45 days after enrollment.
6. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Unlikely to comply with study procedures, restrictions and requirements and judged by the Investigator to be unsuitable for participation.
2. Known pregnancy, per institutional policy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of agreement between I-124 PET and I-123/I-131 SPECT (participant) | 1 day
  Participant-level agreement between I-124 PET and the combination of I-123/I-131 SPECT will be measured. Cohen's kappa will used to measure the level of agreement for individual readers and the consensus read overall, with 95% confidence intervals calculated. A patient will be classified as showing agreement only if all five regions demonstrate agreement; disagreement in one or more regions will result in a classification of disagreement. Additionally, positive and negative percent agreement will be reported with corresponding 95% confidence intervals.
Number of agreement between 1-124 PET and 1-123/1-131 SPECT (region) | 1 day
  Region-level agreement between 1-124 PET and the combination of 1-123/1-131 SPECT will be determined by Individual reader and through a consensus read. A region is in agreement if I-124 PET and I-123/I-131 SPECT results align, either as true positive (both positive) or true negative (both negative). Disagreement occurs when the results diverge, categorized as false positive (I-124 PET positive, but I-123/I-131 SPECT negative) or false negative (I-124 PET negative, but I-123/I-131 SPECT positive).

SECONDARY OUTCOMES:
Overall specificity of I-124 PET to detect metastatic thyroid cancer (participant) | 1 day
  Specificity of I-124 is defined as the proportion of lesions that will be characterized as negative on I-124 PET when compared to the composite truth standard across participants. The composite truth standard is determined by a panel of highly qualified physicians and researchers and will be used to determine true positive (TP), false positive (FP), true negative (TN) and false negative (FN) by participant: o TP: I-124 PET read as positive for tumor, and composite truth standard determined to have tumor. o FP: I-124 PET read as positive for tumor, and composite truth standard determined to not contain tumor. o TN: I-124 PET read as negative for tumor, and composite truth standard determined to not contain tumor. o FN: I-124 PET read as negative for tumor, and composite truth standard determined to contain tumor. Specificity ranges from 0 to 100%, with higher values indicating a better ability for the scan to detect healthy individuals
Overall specificity of I-124 PET to detect metastatic thyroid cancer (region) | 1 day
  Specificity of I-124 is defined as the proportion of lesions that will be characterized as negative on I-124 PET when compared to the composite truth standard by region. The composite truth standard is determined by a panel of highly qualified physicians and researchers and will be used to determine true positive (TP), false positive (FP), true negative (TN) and false negative (FN) by region: o TP: I-124 PET read as positive for tumor, and composite truth standard determined to have tumor. o FP: I-124 PET read as positive for tumor, and composite truth standard determined to not contain tumor. o TN: I-124 PET read as negative for tumor, and composite truth standard determined to not contain tumor. o FN: I-124 PET read as negative for tumor, and composite truth standard determined to contain tumor. Specificity ranges from 0 to 100%, with higher values indicating a better ability for the scan to detect healthy individuals
Overall sensitivity of I-124 PET to detect metastatic thyroid cancer (participant) | 1 day
  Sensitivity of I-124 is defined as the proportion of lesions that will be characterized as positive on I-124 PET when compared to the composite truth standard on a participant level. The composite truth standard is determined by a panel of highly qualified physicians and researchers and will be used to determine true positive (TP), false positive (FP), true negative (TN) and false negative (FN) across participants: o TP: I-124 PET read as positive for tumor, and composite truth standard determined to have tumor. o FP: I-124 PET read as positive for tumor, and composite truth standard determined to not contain tumor. o TN: I-124 PET read as negative for tumor, and composite truth standard determined to not contain tumor. o FN: I-124 PET read as negative for tumor, and composite truth standard determined to contain tumor. Sensitivity ranges from 0 to 100%, with higher values indicating a more sensitive scan.
Overall sensitivity of I-124 PET to detect metastatic thyroid cancer (region) | 1 day
  Sensitivity of I-124 is defined as the proportion of lesions that will be characterized as positive on I-124 PET when compared to the composite truth standard by region. The composite truth standard is determined by a panel of highly qualified physicians and researchers and will be used to determine true positive (TP), false positive (FP), true negative (TN) and false negative (FN) by region: o TP: I-124 PET read as positive for tumor, and composite truth standard determined to have tumor. o FP: I-124 PET read as positive for tumor, and composite truth standard determined to not contain tumor. o TN: I-124 PET read as negative for tumor, and composite truth standard determined to not contain tumor. o FN: I-124 PET read as negative for tumor, and composite truth standard determined to contain tumor. Sensitivity ranges from 0 to 100%, with higher values indicating a more sensitive scan.
Reclassification Rate | 1 day
  Reclassification rate is defined as the proportion of participants what will be characterized as metastatic on I-124 Positron Emission Tomography (PET) that are characterized as localized or nodal only disease on a non-investigational, usual care I-123 Single-photon emission computed tomography (SPECT).
Inter-reader reliability (IRR) for I-124 PET (participant) | 1 day
  Three blinded readers will interpret the non-investigational, usual care I-123 imaging and the I-124 imaging per participants. A Cohen's Kappa will be used to measure the inter-reader variability for I-124 and I-123 separately. Kappa statistics range from -1 to 1 with higher values correspond to higher inter-rater reliability.
Inter-reader reliability (IRR) for I-124 PET (region) | 1 day
  Three blinded readers will interpret the non-investigational, usual care I-123 imaging and the I-124 imaging by region. A Cohen's Kappa will be used to measure the inter-reader variability for I-124 and I-123 separately. Kappa statistics range from -1 to 1 with higher values correspond to higher inter-rater reliability.
Proportion of participants with treatment-related adverse events | Up to 5 days
  Proportion of participants with treatment-related adverse events, as classified and graded by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 5.0).
Proportion of participants with positive I-124 PET in the overall population | 1 day
  The participant level detection rate will be assessed by calculating the number of participants interpreted as having a positive I-124 PET divided by the total number of participants with a scan evaluated by a reader.
Proportion of participants with positive I-124 PET in participants who have negative I-123 SPECT | 1 day
  In the subset of participants where the consensus read of the I-123 imaging study was negative, then the participant level detection rate for this population will be determined. The detection rate will be assessed by calculating the number of participants interpreted as having a positive I-124 PET divided by the total number of participants with a negative I-123 SPECT scan evaluated by a reader.
Mean of total number of lesions characterized as positive on I-124 PET and 24 hour I-123 SPECT | 1 day
  The mean total number of lesions detected for each participant using I-124 and I-123 taken within 24 hours (with a maximum of 10 lesions per region) will be reported along with the variance.
Mean of total number of lesions characterized as positive on both I-124 PET and 7-day post I-131 | 1 day
  The mean total number of lesions detected for each participant using I-124 and I-131 taken within 7 days (with a maximum of 10 lesions per region) will be reported along with the variance.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hope, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No